CLINICAL TRIAL: NCT03593993
Title: A Biospecimen Collection Study to Evaluate the Pharmacokinetic, Pharmacodynamic, and Resistance Profile to Trametinib and Dabrafenib in BRAF-V600E Mutated Recurrent Gliomas
Brief Title: A Biospecimen Collection Study in BRAF-V600E Mutated Recurrent Gliomas
Status: Terminated | Type: Observational
Why Stopped: low accrual and lack of funds
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Musella Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: J1801; IRB00158788 (Other: JHM IRB)
Record Dates: First submitted 2018-06-26; First posted 2018-07-20 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Glioma; BRAF V600E; Pleomorphic Xantho-Astrocytoma; Glioblastoma
MeSH Terms: conditions — Glioma; Astrocytoma; Glioblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, cerebrospinal fluid, tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Surgical Cohort: Blood, cerebrospinal fluid, and tumor tissue will be obtained from each participant on this arm.
  Interventions: Procedure: Surgical Cohort

INTERVENTIONS:
Procedure: Surgical Cohort — Blood, cerebrospinal fluid, and surgical tissue collected during procedure

SUMMARY:
This is a surgical biospecimen collection study. The purpose of this study is to understand how much of two drugs (dabrafenib and trametinib) are able to penetrate brain tumors and turn off the RAF signaling pathway. This is important because these drugs are currently FDA approved for other tumors and may have efficacy in brain tumors with the BRAF V600E mutation.

DETAILED DESCRIPTION:
The primary goal of this study is to establish concentrations of dabrafenib and trametinib in enhancing brain tissue and cerebrospinal fluid from people with BRAF-V600E mutant recurrent gliomas who undergo tumor resection. The exploratory goals are to measure the amount of ERK signaling pathway activity, to identify mechanisms of resistance to these drugs, and evaluate feasibility of measuring tumor DNA in cerebrospinal fluid.

People (adults or children) with brain tumors who are already taking dabrafenib and / or trametinib and are in need of a surgical resection are potentially eligible. On the day of surgery, blood, cerebrospinal fluid, and tumor tissue will be collected for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a history of primary brain tumor (including but not limited to glioblastoma (GBM), anaplastic astrocytoma (AA), anaplastic ganglioglioma (AG), and anaplastic pleomorphic xanthoastrocytoma (PXA)).
* Subjects must have a BRAF-V600 mutation identified in previous tissue analysis (may be IHC or PCR based). Allowable mutations include V600E, V600K, V600R, and V600D.
* Subjects must be taking dabrafenib at a dose of at least 50mg twice daily (adults only) and / or trametinib at a dose of at least 1mg daily (adults only) for at least 7 days prior to surgery as prescribed by their treating physician. Note: Pediatric patients may be taking any dose of dabrafenib and / or trametinib as prescribed by their treating physician for at least 7 days prior to surgery.
* Subjects must be undergoing surgery for clinical purposes.
* Written informed consent - a signed informed consent and/or assent (as age appropriate) for study participation will be obtained according to institutional guidelines.

Exclusion Criteria:

* Subjects who are receiving any other investigational agents or chemotherapeutic agents.
* Subjects for whom collection of blood, spinal fluid, or tissue samples is unsafe or clinically inadvisable.

Min Age: 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary brain tumors who are taking dabrafenib and/or trametinib and are going to have a surgical resection.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2018-05-19 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Concentration of dabrafenib in brain tumor | Day 1
  Obtain single time-point concentration of dabrafenib in enhancing brain tissue (ng/mL) using liquid chromatography/mass spectrometry with one single, random sample
Concentration of trametinib in brain tumor | Day 1
  Obtain single time-point concentration of trametinib in enhancing brain tissue (ng/mL) using liquid chromatography/mass spectrometry with one single, random sample

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Grossman, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Karisa Schreck, MD, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (5):
- United States (5):
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusettes General Hospital, Boston, Massachusetts
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No